CLINICAL TRIAL: NCT00678717
Title: Autonomic Function Testing and Spinal Cord Stimulation: Implications for Successful Therapy in Chronic Visceral Pain
Brief Title: Microneurography and Spinal Cord Stimulation in Chronic Visceral Pain
Acronym: AFTSCSCVP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Peter Konrad, Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 071179
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Chronic Pain
Keywords: abdominal; Pelvic; Pain; SCS; Healthy and Chronic Visceral Pain patients; Chronic Visceral Pain and spinal cord stimulator
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy (Active Comparator): Healthy volunteers
  Interventions: Procedure: Autonomic Evaluation
- Chronic Visceral Pain (Experimental): Chronic Visceral Pain patients. Participants will be tested before and after implantation of a Spinal Cord Stimulator (implantation of the Spinal Cord Stimulator is done as usual care and is not a study procedure)
  Interventions: Procedure: Autonomic Evaluation

INTERVENTIONS:
Procedure: Autonomic Evaluation — Orthostatic vital signs will be determined by measuring heart rate (HR) and brachial blood pressure (BP) during a tilt table test. The degree of vagal mediated sinus arrhythmia will be assessed during controlled breathing (5 seconds inhalation and 5 seconds exhalation during 90 seconds), and the sinus arrhythmia parameters will be calculated as the difference and ratio of the longest to the shortest RR interval. The sympathetic response during breath hold will be measured. Responses of BP, HR, MSNA will be acquired during Valsalva maneuver. The valsalva ratio of heart rate will be calculated from the maximum of heart rate during or shortly after straining and the minimal depressed heart rate in the overshoot phase IV. Blood pressure and MSNA increase during isometric handgrip maintained at 30% of maximal voluntary contraction for five minutes will be determined. The blood pressure and MSNA response will be measured during cold pressor test with the hand in ice water for 1 minute.

SUMMARY:
The purpose of this study is to assess the effect of the spinal cord stimulator (A small wire is surgically implanted under the skin. Low-level electrical signals are then transmitted through the lead to the spinal cord to alleviate pain. Using a magnetic remote control, the patients can turn the current on and off, or adjust the intensity.) on the autonomic nervous system (sympathetic and parasympathetic). Some studies support that the spinal cord stimulation suppresses or decreases sympathetic outflow (the sympathetic nervous system is the one that provide us with the "flight and fight response" and the parasympathetic nervous system is the one that works while we "sleep, rest and digest".). The sympathetic nervous system is important in blood pressure regulation also. However, there are not reports regarding the effect of the spinal cord stimulation on blood pressure regulation in chronic visceral pain patients. Most clinical trials are focus on the effect of the spinal cord stimulation on pain relief. We think we could use blood pressure, heart rate and special analysis of these signals and their relationship to other pain measurements to assess the effect of the spinal cord stimulation in an objective way.

DETAILED DESCRIPTION:
Spinal Cord Stimulation (SCS) has been used since 1967 for the treatment of pain: complex regional pain syndromes 1 , ischemic limb pain 2-5, failed back surgery syndrome 6, 7, and refractory angina pectoris 8-11. Recently, Kapural et al. reported a case series of six patients that underwent SCS for the treatment of chronic visceral pain (CVP)12, 13. SCS reduced 50% of the patients' pain and improved patient functionality by 60% 14 . Animal studies suggested that dorsal column pathways are involved in the transmission of visceral pain 12, 13. Clinical studies in patients with visceral cancer have shown that interruption of the fibers of the dorsal columns that ascend close to the midline of the spinal cord significantly relieves pain and decreases analgesic requirement 15-18. Different studies support the hypothesis that visceral pain perception is positively modulated by the descending pathways from the medulla. Dorsal column lesion leads to a reduction of thalamic activation by visceral stimuli and decreased visceral pain perception 19. Visceral innervation occurs via sympathetic and parasympathetic pathways; parasympathetic afferents enter the vagal afferents carrying nociceptive information enter trunks while sympathetic afferents carrying nociceptive information enter at the levels T6 and L3. Therefore, limited case series using SCS for CVP suggested that pain relief was achieved by blocking these segments suppressing sympathetic outflow to the abdomen and pelvis 14. The relationship between autonomic nervous system (ANS) and pain are poorly understood. Animal and clinical research has provided evidence for close interaction between pain modulatory systems and the ANS 20, 21. However, little is known about the ANS function in chronic pain patients. Our previous funded work suggested that chronic low back pain (CLBP) patients have reduced LFRRI (heart rate variability-low frequency) (not increased as expected) and that indices of the vagal component of the Heart Rate Variability(HRV) (Root Mean Square of the Successive Differences (RMSSD), heart rate variability-high frequency (HFRRI) were also attenuated. The sympatho-vagal balance (LFRRI /HFRRI), a ratio of LF to HF which correlates with higher sympathetic activation 22, was paradoxically increased 23. We previously demonstrated that Low Frequency Systolic Blood Pressure (LFSBP) correlates with muscle sympathetic nerve traffic during orthostatic load supported by a simplified model of blood pressure variability 24. We also showed that LFSBP can be abolished by ganglionic blockade demonstrating the neurogenic origin of these oscillations in blood pressure 25. Additionally, our study revealed decreased baroreflex indices (αHF and BRSLF) during sitting in CLBP patients. Blood pressure was not different in CLBP patients, but there was a trend for higher heart rates possibly caused by higher sympathetic activity to the heart. These findings of reduced baroreflex sensitivity and changes in heart rate support hypothesized alterations in cardio-vagal control in patients with chronic pain 26, 27. In summary, sympathetic function has been assessed by indirect measures. There is no data available regarding the direct assessment of sympathetic outflow in CVP patients. Sympathetic outflow is stimulus specific 28, 29. Therefore, the characterization of resting sympathetic outflow and stimulus-induced sympathetic adjustments requires simultaneous measurements of activity by different techniques. We propose using microneurography to assess the sympathetic function on a second-to-second basis in CVP patients. Microneurography directly assess muscle sympathetic nerve activity (MSNA). This technique is used to define sympathetic responses to a number of standard physiologic maneuvers. It was first developed in Sweden by Wallin, who described the technique for recording afferent muscle or skin sympathetic nerve activity 30, 31. MSNA displays real-time sympathetic nerve activity, allowing definition of sympathetic responses so transient that they would be lost to all other techniques. In general, MSNA burst/min is a good indicator of sympathetic nerve activity 32-37. For example, direct measurement of sympathetic nerve activity as reflected in MSNA has been a very useful tool to demonstrate that increased sympathetic activity is an important factor in the pathogenesis of essential hypertension 38-42. In chronic orthostatic intolerance, a syndrome of autonomic dysfunction in young women MSNA have revealed an abnormal regional distribution of sympathetic activity during orthostatic stress. 43, 44. Moreover, studies in children with complex regional syndrome and adolescents have shown these patients reported systemic ANS symptoms including dizziness, near syncope and postural tachycardia 45-49. Our case series of 5 complex regional pain syndrome patients (4 male, 1 female, 32-51 years) with implanted epidural spinal cord stimulator for pain relief 50 suggested that CRPS (Complex Regional Pain Syndrome) patients have: 1) reduced vasoconstrictor response during Valsalva, 2) A greater blood pressure (BP) drop during straining phase II as compared to normal and less blood pressure overshoot during phase IV in CRPS patients with stimulator turned off and the BP response returns to normal ranges during spinal stimulator turned on. Lastly, muscle sympathetic nerve activity improved during SCS resulting in better blood pressure control. All these data suggest a tight relationship between pain control and sympathetic function. As is well know, CVP is difficult to treat because of its ill-defined nature and treatment with SCS has moderate success, but predicting success in these difficult to treat patients will probably be increased by correlating autonomic function; pain and therapy with spinal cord stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic visceral pain patients candidates for spinal cord stimulation implant with no other chronic diseases.

Exclusion Criteria:

* Diabetes, pulmonary or chronic cardiac diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2009-01-23 (Actual); Study Completion 2009-01-23 (Actual)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity | Prior to stimulator implant and within 1 year of receiving stimulator implant
  Microneurography directly assesses muscle sympathetic nerve activity (MSNA)

SECONDARY OUTCOMES:
Heart rate | Before and up to 1 year after spinal cord stimulator implant
  Participants in both arms will be tested at baseline and again within 1 year. Participants in the Chronic Visceral Pain arm will be tested after implantation of a Spinal Cord Stimulator
blood pressure | Before and up to 1 year after spinal cord stimulator implant
  Participants in both arms will be tested at baseline and again within 1 year. Participants in the Chronic Visceral Pain arm will be tested after implantation of a Spinal Cord Stimulator

CONTACTS AND LOCATIONS:
Overall Officials: Sukdeb Datta, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Interventional Pain Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No